CLINICAL TRIAL: NCT07083297
Title: Study of Readmission to Intensive Care Unit After Cardiac Surgery in Heart Hospital of Assiut University : Risk Factors .Reasons and Early Out Come
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdullah Mohamed sayed Ali, resistant doctor at Assiut university hospital, Assiut University
Other Study IDs: ICU after cardiac surgery
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: patients admitted for cardic surgery

SUMMARY:
Cardiac Surgery is any surgical procedure applied to heart and its connected vessels especially thoracic aorta; representing a treatment option for significant cardiac diseases . As cardiovascular (CVS) diseases is the first leading cause of death worldwide accounting for approximately18 million deaths annually especially in low and middle income countries , medical and surgical treatments are of importance in quality of life of cardiac patient.

Most common causes for cardiac surgery are Coranary artery disease, valvular disease as mitral stenosis or mitral regurgitation, congenital heart diseases. Currently cardiac surgery can provide an advanced treatment for cardiac arrhythmias.

In case of cardiovascular surgery, patient is admitted in Intensive Care Unit (ICU) postoperatively until being stable then discharged. In some cases the patient's state is indicating to be readmitted in ICU, a condition that's required long hospitzation, costs and so, a burden on health services and patient's family.

For controlling this phenomenon; i.e. readmission in ICU, a lot researches were conducted to clarify the leading factors and the outcome in readmitted patients. Preoperative risk factors as renal failure, arrhythmias, chronic obstructive pulmonary disease (COPD) are common noticed factors for readmission of previous heart surgery patient. Also, readmitted patients may have poor clinical outcomes as morbidity and mortality.

In this study we aim to screen for preceding risk factors and report precipitating early events occurring in readmission in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients aged between 18 to 85 years.
* Patients with previous heart surgery.
* Patients will be admitted in Cardiac ICU during the study duration.

Exclusion Criteria:

* Pediatric patients aged below 18 years. b. Elderly Patients aged above 85 years. c. Patient without previous heart surgery. d. Patients are for emergent reoperation. e. Patients admitted in ICU due to Chest Trauma. f. Patients refused consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted for cardic surgery
Sampling Method: Probability Sample
Enrollment: 89 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
mortality rate | 30 day
  mortality rate after cardic surgery